CLINICAL TRIAL: NCT00690482
Title: A 4 Week Double-blind, Placebo-controlled, Randomized, Parallel Group Phase IIa Study to Assess the Efficacy and Safety of AZD1981 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study to Assess the Efficacy and Safety of AZD1981 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Acronym: Columbus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9831C00001
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: Moderate to Severe COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — AZD1981

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1981 (Experimental): AZD1981 Oral tablet, twice daily
  Interventions: Drug: AZD1981
- Placebo (Placebo Comparator): Placebo Oral tablet, twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1981 — Oral tablet, twice daily
  Arms: AZD1981
Drug: Placebo — Placebo Oral tablet, twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to study efficacy and safety of AZD1981 in patients with Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion Criteria:

* FEV1 between 30 and 80% of predicted normal value post-bronchodilator (GOLD stages 2 and 3)
* Clinical diagnosis of COPD

Exclusion Criteria:

* Other clinically relevant disease or disorders
* Exacerbation of COPD within 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jörgen Vestbo, Principal Investigator — Professor in Respiratory Medicine, Hvidovre, Denmark
Locations (21):
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Denmark (4):
  - Research Site, Arhus C
  - Research Site, Hellerup
  - Research Site, Hvidovre
  - Research Site, Værløse
- Poland (5):
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Ostrów Wielkopolski
  - Research Site, Przemyśl
  - Research Site, Rzeszów
- Slovakia (5):
  - Research Site, Bojnice
  - Research Site, Liptovský Hrádok
  - Research Site, Poprad
  - Research Site, Spišská Nová Ves
  - Research Site, Žilina
- Sweden (3):
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uppsala

REFERENCES:
- [Derived] Snell N, Foster M, Vestbo J. Efficacy and safety of AZD1981, a CRTH2 receptor antagonist, in patients with moderate to severe COPD. Respir Med. 2013 Nov;107(11):1722-30. doi: 10.1016/j.rmed.2013.06.006. Epub 2013 Jul 1. PMID 23827726
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=215&filename=CSR-D9831C00001.pdf
- See also: CSR-D9831C00001.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=215&filename=CSR-D9831C00001.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 118 patients were allocated to treatment and 111 completed the study. First patient entered the study on 26 May 2008 and the last patient finished the study on 17 December 2008.
Period: Overall Study
Arm/Group | AZD1981 | Placebo
Started | 61 | 57
Completed | 57 | 54
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Incorrect enrolment | 0 | 1
Not completed — Study-specific discontinuation criteria | 1 | 0
Not completed — Intake of prohibited medicine | 1 | 0
Not completed — withdrew consent at rand.day | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient randomised to placebo withdrew consent immediately after the first dose of investigational product on the day of randomisation. No clinical measurements were performed and no reports of AEs were received for this patient. Since the patient is non-informative both in terms of efficacy and safety, he has been excluded from the analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1981 | Placebo | Total
Number analyzed (Participants) | 61 | 56 | 117
Age, Continuous [Mean (Full Range); unit: Years] | 64.1 [47 to 78] | 62.4 [43 to 83] | 62.4 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: FEV1
Description: Mean change in FEV1 from baseline to Week 4 (last measurement post dose used, if data missing)
Time Frame: Baseline and Week 4
Population: The efficacy analysis is based on 117 randomized patients, 61 on AZD1981 and 56 on placebo. However, not all patients will have valid, non-missing values for a given outcome measure.
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 60 | 55
L | 0.007 (-0.810) [-0.810 to 0.740] | 0.011 (-0.550) [-0.550 to 0.550]

2. Primary Outcome: Clinical COPD Questionnaire
Description: Mean change in Total CCQ from baseline to Week 4 (last measurement post dose used, if data missing). Scores for total CCQ range from 0 (low symptoms) to 6 (high symptoms).
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 59 | 55
Scores on a scale | -0.299 (-2.00) [-2.00 to 1.30] | -0.340 (-2.20) [-2.20 to 1.30]

3. Secondary Outcome: Forced Vital Capacity
Description: Mean change in FVC from baseline to Week 4 (last measurement post dose used, if data missing)
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 60 | 55
L | -0.047 (-1.74) [-1.74 to 0.840] | -0.102 (-1.09) [-1.09 to 0.870]

4. Secondary Outcome: Slow Vital Capacity
Description: Mean change in SVC from baseline to Week 4 (last measurement post dose used, if data missing)
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 60 | 55
L | -0.001 (-1.03) [-1.03 to 2.30] | -0.009 (-1.60) [-1.60 to 0.910]

5. Secondary Outcome: Inspiratory Capacity
Description: Mean change in IC from baseline to Week 4 (last measurement post dose used, if data missing)
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Full Range); unit: L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 60 | 54
L | -0.007 (-0.960) [-0.960 to 1.08] | -0.110 (-1.39) [-1.39 to 1.59]

6. Secondary Outcome: FEF25%-75%
Description: Mean change in FEF25%-75% (forced expiratory flow between 25% and 75% of the FVC) from baseline to Week 4 (last measurement post dose used, if data missing)
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Full Range); unit: L/s
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 60 | 54
L/s | -0.042 (-0.900) [-0.900 to 0.440] | 0.060 (-0.640) [-0.640 to 2.48]

7. Secondary Outcome: COPD Symptom Sleep Score
Description: Mean change in COPD symptom sleep score from baseline to treatment period average (calculated using all available data after randomisation for each patient). Scores for COPD symptom sleep score range from 0 (no symptoms) to 4 (no sleep).
Time Frame: Baseline and 4-week treatment period average
Population: as for outcome 1
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 61 | 56
Scores on a scale | -0.147 (-1.55) [-1.55 to 1.00] | -0.047 (-1.75) [-1.75 to 1.80]

8. Secondary Outcome: COPD Symptom Breathing Score
Description: Mean change in COPD symptom breathing score from baseline to treatment period average (calculated using all available data after randomisation for each patient). Scores for COPD symptom breathing score range from 0 (none) to 4 (severe).
Time Frame: Baseline and 4-week treatment period average
Population: as for outcome 1
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 61 | 56
Scores on a scale | -0.280 (-2.07) [-2.07 to 0.486] | -0.137 (-1.41) [-1.41 to 1.52]

9. Secondary Outcome: COPD Symptom Cough Score
Description: Mean change in COPD symptom cough score from baseline to treatment period average (calculated using all available data after randomisation for each patient). Scores for COPD symptom cough score range from 0 (none) to 4 (almost constant).
Time Frame: Baseline and 4-week treatment period average
Population: as for outcome 1
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 61 | 56
Scores on a scale | -0.202 (-2.09) [-2.09 to 1.22] | -0.124 (-1.79) [-1.79 to 1.01]

10. Secondary Outcome: COPD Symptom Sputum Score
Description: Mean change in COPD symptom sputum score from baseline to treatment period average (calculated using all available data after randomisation for each patient). Scores for COPD symptom sputum score range from 0 (none) to 4 (severe).
Time Frame: Baseline and 4-week treatment period average
Population: as for outcome 1
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 61 | 56
Scores on a scale | -0.300 (-1.50) [-1.50 to 0.844] | -0.290 (-1.58) [-1.58 to 0.796]

11. Secondary Outcome: PEF (Peak Expiratory Flow) Morning
Description: Mean change in PEF morning from baseline to treatment period average (calculated using all available data after randomisation for each patient).
Time Frame: Baseline and 4-week treatment period average
Population: as for outcome 1
Measure: Mean (Full Range); unit: L/min
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 61 | 56
L/min | 2.86 (-45.0) [-45.0 to 113] | 4.54 (-37.2) [-37.2 to 77.9]

12. Secondary Outcome: PEF (Peak Expiratory Flow) Evening
Description: Mean change in PEF evening from baseline to treatment period average (calculated using all available data after randomisation for each patient).
Time Frame: Baseline and 4-week treatment period average
Population: as for outcome 1
Measure: Mean (Full Range); unit: L/min
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 60 | 56
L/min | -1.61 (-66.5) [-66.5 to 115] | 5.73 (-35.1) [-35.1 to 61.8]

13. Secondary Outcome: Total Use of Reliever
Description: Mean change in Total use of reliever from baseline to treatment period average (calculated using all available data after randomisation for each patient).
Time Frame: Baseline and 4-week treatment period average
Population: as for outcome 1
Measure: Mean (Full Range); unit: Number of inhalations per day
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 59 | 55
Number of inhalations per day | -0.330 (-7.64) [-7.64 to 3.81] | -0.139 (-3.69) [-3.69 to 9.90]

14. Secondary Outcome: Adverse Event
Description: The number of participants that experienced at least one adverse event.
Time Frame: Up to 4 Weeks
Population: The safety analysis is based on 117 randomized patients, 61 on AZD1981 and 56 on placebo.
Measure: Number; unit: Participants
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 61 | 56
Participants | 20 | 18

ADVERSE EVENTS:
Arm/Group | AZD1981 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/61 | 1/56
Other Adverse Events (participants affected / at risk) | 8/61 | 6/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1981 (N=61) | Placebo (N=56)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1981 (N=61) | Placebo (N=56)
NASOPHARYNGITIS (Infections and infestations) | 6 | 3
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less